CLINICAL TRIAL: NCT05080556
Title: A Multicentre Phase II Randomised Controlled Trial to Evaluate the Efficacy of Adaptive Therapy (AT) With Carboplatin, Based on Changes in CA125, in Patients With Relapsed Platinum-sensitive High Grade Serous or High Grade Endometrioid Ovarian Cancer
Brief Title: Adaptive ChemoTherapy for Ovarian Cancer in Patients With Replased Platinum-sensitive High Grade Serous or High Grade Endometrioid Ovarian Cancer
Acronym: ACTOv
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Anticancer Fund, Belgium (Other); JP Moulton Charitable Foundation (Other); Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 136618
Record Dates: First submitted 2021-06-16; First posted 2021-10-15 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer; Relapsed Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Endometrioid Carcinoma; High Grade Serous Carcinoma; Ovary Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Endometrioid | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (control) - standard dosing carboplatin (Active Comparator): Arm 1 (Standard Dosing): Carboplatin AUC5 based on nuclear medicine renal clearance.
  Interventions: Drug: Carboplatin
- Arm 2 (experimental) - adaptive therapy carboplatin according to CA125 (Experimental): Arm 2 (Adaptive Therapy): Carboplatin dose will be calculated according to the CA125 value.
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Carboplatin — Treatment in both arms will be administered intravenously (IV) every 21 days (q21D) and for a maximum of 6 cycles in Arm 1 and 12 cycles in Arm 2.

SUMMARY:
ACTOv will compare standard 3-weekly carboplatin (AUC5), to carboplatin delivered according to an AT regimen. The AT regimen will modify carboplatin dose according to changes in the clinical-standard serum biomarker CA125 as a proxy measure of total tumour burden and an individual patient's response to the most recent chemotherapy treatment. AT could prolong sensitivity to carboplatin and extend tumour control, while simultaneously reducing chemotherapy dose and drug-induced toxicity. Carboplatin is a low cost and low toxicity drug that has an enduring and central role in ovarian cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years
2. ECOG performance status 0-2
3. Histologically proven diagnosis of high grade serous or high grade endometrioid carcinoma of the ovary, fallopian tube or peritoneum
4. Most recent regimen must have included platinum (cisplatin or carboplatin)
5. Must have previously received a PARP inhibitor
6. 6. Must have responded to most recent platinum treatment by CT or MRI or by GCIG CA125 response criteria
7. Pre-trial CT or MRI-confirmed disease relapse ≥ 6 months after day 1 of the last cycle of platinum-containing chemotherapy (cisplatin or carboplatin) and requiring treatment with further platinum-based chemotherapy
8. Measurable disease by RECIST v1.1 on a CT scan conducted within 28 days prior to randomisation (Patient with non-measurable disease could be eligible if they meet GCIG CA125 progression criteria)
9. CA125 ≥ 100iU/l at screening
10. Agree to provide additional research blood samples at the same time as blood draws prior to each carboplatin treatment, 6-weekly during surveillance and at 12- weekly follow-up visit
11. Expected to be able to commence treatment within 28 days post randomisation
12. Adequate bone marrow function
13. Adequate liver function
14. Adequate renal function
15. Postmenopausal or women of child-bearing potential (WOCBP) must agree to have an urine or serum pregnancy test at screening for evidence of non-childbearing status and prior to trial treatment and use adequate contraception for duration of trial
16. Willing and able to give consent and able to comply with treatment and follow up schedule

Exclusion Criteria:

1. Non-epithelial ovarian cancer, carcinosarcoma, low-grade serous and endometrioid carcinomas, mucinous & clear-cell carcinomas
2. Patients requiring treatment with combination chemotherapy regimens
3. Patients with a known hypersensitivity to carboplatin
4. Persisting ≥ grade 2 CTCAE v5 adverse events/ toxicity (except alopecia and neuropathy) from previous anti-cancer treatment.
5. Treatment with any other investigational agent, or participation in another interventional clinical trial within 28 days prior to randomisation.
6. Major surgery within 14 days before anticipated start of treatment and patients must have recovered from any effects of major surgery.
7. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicated the use of an investigation drug or puts the patients at high risk for treatment-related complications.
8. Other psychological, psychiatric, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
9. Malignancy treated within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, Stage 1, grade 1 endometrial carcinoma.
10. Patients with symptomatic uncontrolled brain or meningeal metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
11. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days prior to randomisation.
12. Pregnant or breast-feeding women are excluded. Women of childbearing potential will be excluded unless effective methods of contraception are used from signing of the informed consent, throughout the period of taking study treatment and for at least 6 months after last dose of trial drug(s).
13. Inability to attend or comply with treatment or follow-up scheduling.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Modified Progression Free Survival (mPFS) | From the date of randomisation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years.
  Measured from the date of randomisation to the date of objective progression (investigator assessed using RECIST v1.1) but comparing CT scans to the baseline CT rather than the radiological nadir), clinical progression or death from any cause (in the absence of progression)

SECONDARY OUTCOMES:
Acceptability (1/2) | From the date of randomisation to the first dose of treatment (within 28 days from randomisation)received by patient. Measured as the number of patients approached who accept randomisation.
  the number of eligible patients approached who accept randomisation and continue to receive treatment
Acceptability (2/2) | From the date of randomisation to the first dose of treatment (within 28 days from randomisation)received by patient. Measured as the percent of patients approached who accept randomisation.
  the proportion of eligible patients approached who accept randomisation and continue to receive treatment
Deliverability (1/2) | Measured as the number of treatment cycles that are delivered as per protocol, described by trial arm (maximum of 6 cycles in control arm and 12 in experimental arm, approx.. 18 weeks and 36 weeks respectively). Treatment delays, reductions and omissions
  the number of treatment cycles that are delivered as per protocol, described by trial arm
Deliverability (2/2) | Measured as the number of treatment cycles that are delivered as per protocol, described by trial arm (maximum of 6 cycles in control arm and 12 in experimental arm, approx.. 18 weeks and 36 weeks respectively). Treatment delays, reductions and omissions
  the proportion of treatment cycles that are delivered as per protocol, described by trial arm
Compliance | Total cumulative carboplatin dose will be calculated for each patient over time on treatment (max. of 6 cycles in control arm and 12 cycles in experimental arm, approximately 18 weeks and 36 weeks respectively
  total cumulative carboplatin dose will be calculated for each patient over time on treatment, and described by trial arm
Adverse events (1/2) | Adverse events will be reported between informed consent and 30 calendar days post last IMP (i.e. max. of 6 cycles in control arm and 12 cycles in experimental arm, approximately 30 days after 18 weeks or 36 weeks respectively)
  adverse events will be categorised using the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5. The number of patients who suffer a grade 3 or 4 toxicity at any time, and the maximum grade of toxicity for each adverse event term, will be described by trial arm
Adverse events (2/2) | Adverse events will be reported between informed consent and 30 calendar days post last IMP (i.e. max. of 6 cycles in control arm and 12 cycles in experimental arm, approximately 30 days after 18 weeks or 36 weeks respectively)
  adverse events will be categorised using the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5. The percentage of patients who suffer a grade 3 or 4 toxicity at any time, and the maximum grade of toxicity for each adverse event term, will be described by trial arm
Quality of life (1/2) - EORTC questionnaire (assessing the quality of life of patients with ovarian cancer) | At baseline, during treatment and follow up until the first documented progression or date of death (estimate 6 or 12 months but can be up to 4 years)
  measured using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC questionnaires): Quality of Life cancer 30 (QLQ-C30) (suitable for all cancer types) and Qualify of life questionnaire (QLQ-OV28 (ovarian cancer-specific)) in scale of 4 (1 is not very much and 4 very much)
Quality of life (2/2) - EQ-5D ((mobility, self-care, usual activities, pain/discomfort, anxiety/depression, a single summary index and a visual analogue scale) | At baseline, during treatment and follow up until the first documented progression or date of death (estimate 6 or 12 months but can be up to 4 years)
  measured using European Quality of life questionnaire five dimensions (EQ-5D (descriptive profile of health state)) in scale of 5 (1 is no problem and 5 is extreme problem)
Fear of progression | At baseline, during treatment and follow up until the first documented progression or date of death (estimate 6 or 12 months but can be up to 4 years)
  measured using Fear of progression questionnaire (FOP-Q SF) in scale of 1 to 5 where 1 is never and 5 is very often
CA125 | Measured at baseline, 3 weekly during treatment, 6-weekly during surveillance and 12-weekly during follow-up, through study completion, an average of 1 year.
  measured at baseline, 3-weekly during treatment, 6-weekly during surveillance and 12-weekly during follow-up
Further treatment (1/3) | Additional treatment of patients who progress will be described by trial arm, this will include the time-to-next treatment (measured from randomisation).
  of patients who progress will be described by trial arm including the time-to-next treatment (measured from randomisation)
Further treatment (2/3) | Additional treatment of patients who progress will be described by trial arm, this will include the time treatment received (measured from randomisation)
  of patients who progress will be described by trial arm including the time treatment received (measured from randomisation)
Further treatment (3/3) | Additional treatment of patients who progress will be described by trial arm, this will include the time response to this treatment (measured from randomisation)
  of patients who progress will be described by trial arm including the time response to this treatment (measured from randomisation)
Overall survival | Measured from the date of randomisation to the date of death from any cause, censored at the date last seen (estimate 2 years but can be up to 4 years)
  measured from the date of randomisation to the date of death from any cause. Patients who are event-free will be censored at the date last seen

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals, London, United Kingdom

REFERENCES:
- [Derived] Mukherjee UA, Hockings H, Counsell N, Patel A, Narayanan P, Wilkinson K, Dhanda H, Robinson K, McNeish I, Anderson ARA, Miller R, Gourley C, Graham T, Lockley M. Study protocol for Adaptive ChemoTherapy for Ovarian cancer (ACTOv): a multicentre phase II randomised controlled trial to evaluate the efficacy of adaptive therapy (AT) with carboplatin, based on changes in CA125, in patients with relapsed platinum-sensitive high-grade serous or high-grade endometrioid ovarian cancer. BMJ Open. 2024 Dec 22;14(12):e091262. doi: 10.1136/bmjopen-2024-091262. PMID 39806715